



# Participant Informed Consent Form (ICF)

Balanced Progressive Intensity Training (BPIT) Multi-Site Clinical Study Version 1.1

MMSx Authority Institute for Movement Mechanics & Biomechanics Research In Collaboration with BodyGNTX Institute | GFFI India | IIKBS | Bureau of Fitness Standards (BFS) | Active India Health & Fitness Trust (AIHFT)

"Note: This latest ICF doc is approved by MMSx Authority Ethics Committee on November 24, 2025"

Date: November 24, 2025

#### **Version History:**

- Version 1.0: Initial draft, November 6, 2025.
- Version 1.1: Reviewed for ClinicalTrials.gov submission on November 24, 2025; no changes to consent procedures or risks.

## 1. Study Title

**Balanced Progressive Intensity Training (BPIT):** A Multi-Site Clinical Evaluation of Movement Efficiency, Mobility, and Strength Adaptation in Healthy Adults (18-65 years).

## 2. Purpose of the Study

You are invited to participate in a **5-week clinical study** that evaluates the effects of the **BPIT method** on movement efficiency, joint mobility, postural alignment, and strength performance. The purpose is to understand how the **BPIT 5-Line Principle** improves biomechanical safety, neuromuscular activation, and training outcomes in healthy individuals.

## 3. Procedures

If you agree to participate, the following procedures will be carried out over the 5-week study duration:

- You will undergo baseline biomechanical screening and mobility testing.
- You will perform training sessions following the BPIT framework under MMSx-certified experts for **5 weeks**.





- Your weekly progress will be documented, including pain scales, posture, range of motion, and strength outcomes.
- Data from this study (anonymized, no personal identifiers) may be used in a U.S. university dissertation under co-IRB oversight, ensuring privacy and ethical review.

If at any time you experience **discomfort**, **pain**, **or fatigue**, you should immediately inform your instructor or clinical supervisor.

#### 4. Potential Risks and Discomforts

Participation in physical activity involves minimal risk, such as:

- Temporary muscle soreness or fatigue.
- Mild joint stiffness or discomfort.
- In rare cases, aggravation of pre-existing injuries.

To minimize these risks, all sessions are supervised by qualified professionals, and the BPIT protocol is **individualized** based on each participant's capacity.

### 5. Benefits

Participation in this study may improve:

- Posture and movement efficiency.
- Strength and endurance.
- Joint mobility and balance.
- Understanding of personal biomechanics and recovery needs.
- As compensation, participants receive free BPIT training sessions (valued at \$100) and a completion certificate for personal records.

Results from this study may help create safer and more effective strength-training methods for athletes and the general population.

## 6. Confidentiality

All data collected will remain **confidential** and used solely for scientific analysis and improvement of training safety protocols.

- All personal information will be coded and kept confidential within the BodyGNTX Research Registry.
- Your identity will **not** appear in any report, publication, or presentation related to this study.
- Data will be stored securely for academic and clinical purposes only.

## 7. Voluntary Participation and Withdrawal

Participation is voluntary.





- You may choose not to participate or withdraw at any time without penalty or loss of benefits.
- If you withdraw, no further data will be collected from you. Previously collected data will remain securely stored for institutional integrity records.

# 8. Medical Oversight and Emergency Protocol

- **Medical professionals** (orthopedists, physiotherapists, and sports physicians) are available at each study site.
- In the event of any injury or health event, appropriate **medical attention will be provided immediately**.
- All adverse events must be documented in the Observation Log and reported to the MMSx Clinical Oversight Board.

## 9. Contact Information

For questions regarding the study, you may contact:

| 1 5 5 | , | |
|---|---|---|
| Role | Name | Contact |
| Principal Investigator | Dr. Neeraj Mehta, Ph.D. | Email: |
| | | info@mmsxauthority.com |
| Institute | MMSx Authority Institute for | |
| | Movement Mechanics & | |
| | Biomechanics Research | |

## 10. Consent Statement

I have read and understood the above information. I voluntarily agree to participate in this study under the supervision of the MMSx research and training team. I understand that I may withdraw at any time without giving a reason, and that my data will be kept confidential.

## **Participant Declaration**

| Field | Entry | Field | Entry |
|-----------------------|-------|----------------|-------|
| Participant Name | | Contact Number | |
| Participant Signature | | Date | |

## **Investigator Declaration**

I have explained the study details to the participant in a clear and understandable manner. All questions have been answered truthfully to ensure informed participation.





| Field | Entry | Field | Entry |
|------------------------|-----------------|-----------|-------|
| Investigator Name | Principle | Signature | |
| Principle Investigator | Dr Neeraj Mehta | Shaha | |
| Site Investigator | | | |
| Designation / Site | | Date | |

## Witness (Optional)

| Name | Signature | Date |
|------|-----------|------|

© 2025 MMSx Authority Institute for Movement Mechanics & Biomechanics Research In Collaboration with BodyGNTX | GFFI India | IIKBS | BFS | AIHFT IMSO Accreditation ID: Appendix A: Bilingual Informed Consent (English/Hindi)

Official: English. Hindi for India sites (GFFI/BFS/AIHFT). Contact PI for questions. (BPIT v3.2 Nov 24, 2025)

## English (Official)

1. Study Title BPIT: Multi-Site Eval of Movement Efficiency, Mobility & Strength in Adults (18-52 yrs).

#### Hindi Translation

1. अध्ययन शीर्षक BPIT: वयस्कों (18-52 yrs) में गति दक्षता, गतिशीलता & शक्ति का बह-साइट मूल्यांकन।





- **2. Purpose** 5-week study evaluates BPIT effects on efficiency, mobility, alignment, strength. Understands 5-Line Principle for safety, activation, outcomes in healthy people.
  - गतिशीलता, संरेखण, शक्ति पर प्रभावों का tivation, मूल्यांकन। 5-लाइन सिद्धांत से सुरक्षा, सक्रियण, परिणामों को समझना।
- 3. Procedures Over 5 weeks: Baseline screening/testing; BPIT sessions (MMSx experts); Weekly docs (pain, posture, ROM, strength). Report discomfort immediately. Anonymized data may use in U.S. dissertation (co-IRB, privacy ensured).
- 3. प्रक्रियाएँ 5 सप्ताह में: बेसलाइन स्क्रीनिंग/परीक्षण; BPIT सत्र (MMSx विशेषज्ञ); साप्ताहिक दस्तावेज (दर्द, मुद्रा, ROM, शक्ति)। असुविधा तुरंत रिपोर्ट करें। गुमनाम डेटा U.S. शोध प्रबंध में उपयोग (सह-आईआरबी, गोपनीयता सुनिश्चित)।

2. उद्देश्य 5-सप्ताह अध्ययन BPIT के दक्षता.

- **4. Risks** Minimal: Temporary soreness/fatigue; mild stiffness; rare injury aggravation. Minimized by supervision & individualized protocol.
- 4. जोखिम न्यूनतमः अस्थायी दर्द/थकानः; हल्की कठोरताः; दुर्लभ चोट बिगड़ना। पर्यवेक्षण & व्यक्तिगत प्रोटोकॉल से कम।
- **5. Benefits** May improve efficiency/mobility, alignment/strength, safety/outcomes. Compensation: Free BPIT sessions (\$100 value) + completion cert.
- 5. लाभ दक्षता/गतिशीलता, संरेखण/शक्ति, सुरक्षा/परिणाम सुधार। मुआवजा: मुफ्त BPIT सत्र (\$100 मूल्य) + पूर्णता प्रमाणपत्र।